CLINICAL TRIAL: NCT05553210
Title: Effects of Intervention Plan on Outcomes of Stress Recovery Program FOREST+ for Healthcare Workers: A Randomized Controlled Trial
Brief Title: Internet-Based Stress Recovery Program FOREST+ for Healthcare Workers
Acronym: FOREST+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25 / (1.3) 250000-KP-22-III
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2022-09

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Forests

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated either to the intervention or control groups. The intervention group will use the intervention with an intervention plan and the control - without an intervention plan. Both groups will participate in the program at the same time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a 6-week therapist-guided online stress recovery intervention with an intervention plan.
  Interventions: Behavioral: FOREST+
- Control group (Experimental): The control group will get a 6-week therapist-guided online stress recovery intervention without an intervention plan. The control group will participate in the program at the same time as the intervention group.
  Interventions: Behavioral: FOREST+

INTERVENTIONS:
Behavioral: FOREST+ — The intervention will be delivered as an internet-based stress recovery intervention consisting of six weekly modules: introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. Each module consists of a psychoeducational and an exercise component. During the program, a therapist provides individual feedback on the completed exercises and can also be available on request.

SUMMARY:
The study aims to assess the efficacy of an internet-based stress recovery intervention for healthcare workers receiving therapist support with or without an intervention plan.

DETAILED DESCRIPTION:
The intervention will be delivered as an internet-based stress recovery program for healthcare workers, comprising of six modules: introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. These modules have been chosen after considering themes that could be most useful for healthcare workers under high stress. Each module consists of a psychoeducational and an exercise component. An intervention plan will be drawn up with the therapist prior to the start of the program, setting the intensity of engagement and the frequency of reminders. During the program, a therapist provides individual feedback on the completed exercises and can also be available on request.

The effect of the intervention will be compared with a control group that will use the program without an intervention plan. The intervention will be delivered in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* licensed healthcare professionals currently working under license;
* at least 18 years old;
* comprehending Lithuanian language;
* access to internet.

Exclusion Criteria:

* acute psychiatric crisis;
* high suicide risk;
* interpersonal violence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change on Recovery Experience Questionnaire | Pre-treatment, post-treatment (after 6 weeks), 6 months follow-up
  Changes on stress recovery are measured. Recovery Experiences Questionnaire (Sonnentag & Fritz, 2007) is a selfreport measure consisting of 16 questions. All items are answered on a 5-point Likert scale ranging from 1 (Totally disagree) to 5 (Totally agree). A higher score indicates more pronounced recovery.

SECONDARY OUTCOMES:
Change on Perceived Stress Scale | Pre-treatment, post-treatment (after 6 weeks), 6 months follow-up
  Changes on perceived stress are measured. Perceived Stress Scale (PSS-4, Cohen et al., 1983) is a self-report measure and consists of 4 questions. All items are answered on a 5 point Likert scale that ranges from 0 (Never) to 4 (Very often). Higher score indicates more pronounced perceived stress.
Change on Patient Health Questionnaire | Pre-treatment, post-treatment (after 6 weeks), 6 months follow-up
  Changes on anxiety and depression symptoms are measured. Patient Health Questionnaire-4 (PHQ-4, Kroenke et al., 2001) is a self-report measure and consists of 4 questions. All items are answered on a 4-point Likert scale that ranges from 0 (Not at all) to 3 (Nearly every day). Higher score indicates more pronounced anxiety or depression symptoms.
Change on Well-being Index | Pre-treatment, post-treatment (after 6 weeks), 6 months follow-up
  Changes on well-being are measured. Well-being Index (WHO-5, Bech, 2004) is a self-report measure and consists of 5 questions. All items are answered on a 6-point Likert scale that ranges from 0 (At no time) to 5 (All of the time). Higher score indicates more pronounced well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Kazlauskas, Ph.D., Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nomeikaite A, Gelezelyte O, Bottche M, Andersson G, Kazlauskas E. Role of Tailored Timing and Frequency Prompts on the Efficacy of an Internet-Delivered Stress Recovery Intervention for Health Care Workers: Randomized Controlled Trial. JMIR Ment Health. 2025 Jan 28;12:e62782. doi: 10.2196/62782. PMID 39874572